CLINICAL TRIAL: NCT03248752
Title: Physical Activity Promotion Through Wearable Monitors: A Test of Self and Partner Monitoring Strategies.
Brief Title: Monitoring Physical Activity (Fitbit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, Principal Investigator, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BC17-180
Record Dates: First submitted 2017-07-26; First posted 2017-08-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2018-11

CONDITIONS: Physical Activity; Health Promotion
Keywords: Behavioural
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Self monitored (Active Comparator): Fitbit use and reports details: Participants will receive a Fitbit device to wear for 3 months. They will engage with the Fitbit application on their smartphone or tablet device and receive a Weekly Progress Report from Fitbit.
  Interventions: Behavioral: Fitbit use and reports
- Group 2 - Partner monitored (Experimental): Fitbit use and reports details: Participant will receive a Fitbit device to wear for 3 months. They will engage with the Fitbit application on their smartphone or tablet device. Participant will also engage with their partner through the Fitbit application. They will have access to their partner's daily progress and be able to communicate through the application. They will also receive their partner's Weekly Fitbit Reports and have a weekly discussion about the Weekly Fitbit Report.
  Interventions: Behavioral: Fitbit use and reports; Behavioral: Partner engagement

INTERVENTIONS:
Behavioral: Fitbit use and reports — Participants will receive a Fitbit device to be used for the duration of the study. Participants will engage with the Fitbit and application and receive Weekly Progress Reports from Fitbit.
Behavioral: Partner engagement — Participants will be connected with their partner in the Fitbit app and therefore have the ability to access their partner's progress. Participants' Weekly Progress Reports will be automatically forwarded to their partner. Participants will engage in a weekly discussion on the topic of their Weekly Progress Reports.
  Arms: Group 2 - Partner monitored

SUMMARY:
The purpose of this study is to examine the effect of monitoring and sharing physical activity outcomes (using Fitbit technology) with a domestic partner on physical activity participation.

Primary research question: Does sharing physical activity outcomes from wearable technology with a participant's partner improve overall physical activity over 3 months compared to not sharing outcomes? Physical activity will be measured as minutes of moderate to vigorous physical activity per week.

Hypothesis: Knowledge that physical activity outcomes are visible to a participant's partner will serve as a proxy-supervision intervention. Awareness of partner's progress will serve as further motivation. Both factors will improve physical activity adherence in comparison to participants without shared outcomes.

DETAILED DESCRIPTION:
Background: Physical activity is associated with management and/or prevention of over 25 chronic health conditions; however the majority of adults in North America are not active enough to experience these benefits. Behavioral strategies have been shown to be effective for increasing physical activity, and wearable fitness monitors such as Fitbits include components of several behavioral strategies including goal setting and feedback. While this technology provides a platform for implementing self-regulation techniques important for behavior change, direct supervision is still the most effective strategy for behavior change. Supervised exercise programs and personal trainers may not be accessible or affordable for people; this study will examine whether proxy supervision by a partner is effective in changing behavior compared to self-regulation alone.

Target Population: Sedentary adults aged 45-75 years old living in Victoria, British-Columbia, Canada.

Sample Size: 80 participant pairs (160 total participants), 40 pairs per group (80 participants per group).

Intervention: Participants will be randomized to two groups: 1 - Self Monitored, 2 - Partner monitored. Both groups will receive an intervention with Group 1 (Self monitored) serving as the comparison group. Participants from both groups will wear an accelerometer for 1 week and complete an online questionnaire at baseline, 6 weeks, and 3 months. Measures of height, weight, waist circumference, and resting blood pressure and heart rate will be taken at baseline and 3 months. Participants will all receive a Fitbit activity tracker and wear it for 3 months. Group 2 (Partner monitor) participants will also have access to their partner's daily progress, receive eachother's Weekly Fitbit reports, and engage in a weekly discussion related to their Weekly Fitbit Report.

ELIGIBILITY:
Inclusion Criteria:

* One or both partners currently not meeting the Canadian Physical Activity Guidelines of 150 minutes of moderate to vigorous physical activity per week
* Currently living in Victoria, BC
* Safe to participate in physical activity (physician clearance required if applicable)

Exclusion Criteria:

* No smartphone or tablet device (with bluetooth technology)
* No email address
* No partner and/or not living with partner

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in participants' weekly physical activity participation at 3 months. | Baseline, 6 weeks, and 3 months
  Quantified as minutes of moderate to vigorous physical activity measured with accelerometry. Participants will wear an accelerometer for a minimum of 10 hours per day for 7 consecutive days. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).

SECONDARY OUTCOMES:
Change in Body Mass Index from baseline to 3 months. | Baseline and 3 months
  Standardized protocols for measuring weight in kilograms (kg) and height in centimeters (cm) will be performed as per the Canadian Society for Exercise Physiology guidelines. Body Mass Index (BMI) will be calculated as kg/m^2. Body Mass Index is an indicator of body composition which is associated with physical activity. Changes in BMI will be examined (3 months to baseline).
Change in waist circumference from baseline to 3 months. | Baseline, 3 months
  Standardized protocols for measuring waist circumference in centimeters (cm) will be performed as per the Canadian Society for Exercise Physiology guidelines. Waist circumference is an indicator of body composition which is associated with physical activity. Changes in waist circumference will be examined (3 months to baseline).
Change in self-reported physical activity from baseline to 3 months. | Baseline, 6 weeks, 3 months.
  Measured from questionnaire using Godin's personal self report leisure time measurement tool, also known as the Leisure Score Index (LSI). The Leisure Score Index contains three questions, which assess the frequency of mild, moderate, and strenuous activity performed for at least 15 minutes during free time in a typical week. Changes in these measures will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in quality of life from baseline to 3 months measured using the Short Form 12 questionnaire. | Baseline, 6 weeks, 3 months
  The online questionnaire will asses participants' quality of life using the short form 12 questionnaire. Changes in this measures will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in life satisfaction from baseline to 3 months measured using Diener's satisfaction with life scale in a questionnaire. | Baseline, 6 weeks, 3 months
  The online questionnaire will asses participants' life satisfaction using Diener's satisfaction with life scale. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in mood from baseline to 3 months measured using the Hospital Anxiety and Depression Scale in a questionnaire. | Baseline, 6 weeks, 3 months
  The online questionnaire will asses participants' mood using the Hospital Anxiety and Depression scale. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in physical activity beliefs, attitudes, barriers, and motivation from baseline to 3 months. | Baseline, 6 weeks, 3 months
  Included in questionnaire - Ajzen's theory of planned behaviour questionnaire will be applied to measure participants' beliefs, attitudes, barriers, and motivation related to physical activity. Changes in these measures will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in physical activity behaviour regulation from baseline to 3 months. | Baseline, 6 weeks, 3 months
  Included in questionnaire - 5 items adapted from Umstattd's scale measuring physical activity self-regulation strategies in older adults. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in physical activity habits from baseline to 3 months. | Baseline, 6 weeks, 3 months
  Included in questionnaire - 12 Self Report Habit Index items from the measure developed by Verplanken and Orbell and adapted to physical activity by Chatzisarantis and Hagger. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).
Change in physical activity identity from baseline to 3 months. | Baseline, 6 weeks, 3 months
  Included in questionnaire - Anderson and Cychosz Exercise Identity Scale is used to measure participants' identification as someone who participates in physical activity. Changes in this measure will be examined (3 months to baseline, 3 months to 6 weeks, 6 weeks to baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Scott Hofer, PhD, Study Chair — University of Victoria
Locations (1):
- Behavioural Medicine Lab, University of Victoria, Victoria, British Columbia, Canada